CLINICAL TRIAL: NCT05021068
Title: Investigation of The Relationship Between Spinal Structure and Mobility and Respiratory Functions in Chronic Obstructive Pulmonary Disease
Brief Title: Spinal Structure and Mobility in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: IKC1233
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: COPD; Postural; Defect; Respiratory Function Impaired; Dyspnea
Keywords: copd; posture; respiratory function; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Dyspnea; Respiratory Aspiration | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD Patients: The respiratory functions of the participants will be measured in accordance with the ATS-ERS criteria. After measurement; forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC, total lung capacity (TLC), residual volume (RV), inspiratory capacity (IC), vital capacity (VC) parameters will be recorded.
  Spinal structure and mobility will be evaluated with the Spinal Mouse device in the sagittal and frontal planes in standing and sitting positions. For the sagittal plane, the measurements were first in the neutral, then in the maximum flexion and extension positions, for the frontal plane; neutral, right and left lateral flexions will be performed.
  Patients will be asked to mark the level of activity that causes dyspnea on the Medical Council Research Scale (MMRC) Dyspnea Score.
  Interventions: Other: Postural Assessment
- Control Group: The respiratory functions of the participants will be measured in accordance with the ATS-ERS criteria. After measurement; forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC, total lung capacity (TLC), residual volume (RV), inspiratory capacity (IC), vital capacity (VC) parameters will be recorded.
  Spinal structure and mobility will be evaluated with the Spinal Mouse device in the sagittal and frontal planes in standing and sitting positions. For the sagittal plane, the measurements were first in the neutral, then in the maximum flexion and extension positions, for the frontal plane; neutral, right and left lateral flexions will be performed.
  Patients will be asked to mark the level of activity that causes dyspnea on the Medical Council Research Scale (MMRC) Dyspnea Score.
  Interventions: Other: Postural Assessment

INTERVENTIONS:
Other: Postural Assessment — Spinal mouse measurement
  Other Names: Respiratory Function Test; MMRC Dyspnea measurement

SUMMARY:
In recent studies with musculoskeletal system disorders in chronic respiratory patients, it has been reported that postural control is affected in COPD patients.

The aim of this study to investigate relationship between spinal structure and mobility an severity of dyspnea in patients with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a preventable and treatable disease characterized by irreversible airway limitation. In recent studies with musculoskeletal system disorders in chronic respiratory patients, it has been reported that postural control is affected in COPD patients.It has been observed that balance systems, functional balance tests, posturography, posture assessment systems, force platform and inclinometer measurements are used in studies on postural control assessment in COPD patients.There are a limited number of studies in which devices that objectively present the degree of deviation in spinal curves are used in patients with COPD, and posture and lung volume and capacities are evaluated.

Therefore, the aim of this study is to investigate the changes in spine structure and mobility in COPD patients and to reveal their relationship with static and dynamic lung volumes and capacities.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Be over 18 years old
* Being clinically stable
* Not having a COPD attack in the last 3 months at least

Exclusion Criteria:

* Refusing to participate in the research
* Having had spinal surgery Presence of back and shoulder pain
* Idiopathic scoliosis
* Ankylosing spondylitis
* Presence of respiratory disease other than COPD
* Difficulty understanding verbal commands

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Spinal Structure and Mobility | 15 minutes (single application)
  Spinal mouse measurement

SECONDARY OUTCOMES:
Pulmonary Functions | 10 minutes (single application)
  Respiratory Function Test
Dyspnea Severity | 5 minutes (single application)
  Modified Medical Research Dyspnea Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No